CLINICAL TRIAL: NCT00819078
Title: Randomized, Double-Blind, Placebo-Controlled Trial of SR Bupropion for Adolescent Smoking Cessation
Brief Title: Comparative Study of SR Bupropion for Adolescent Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Geha Mental Health Center (Other)
Responsible Party: Dr. Gal Shoval, Geha Meantal Health Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GehaMHC; No grants so far
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Smoking; Smoking Cessation
Keywords: adolescent; bupropion; smoking; cessation; depression
MeSH Terms: conditions — Smoking; Smoking Cessation; Depression | interventions — Bupropion; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupropion Sr (Active Comparator): 40 adolescent patients
  Interventions: Drug: Bupropion
- Placebo (sugar pill) (Placebo Comparator): 40 adolescent patients will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupropion — 300 mg/d
  Arms: Bupropion Sr
Drug: Placebo — no dosage
  Other Names: Sugar pill serving as placebo
  Arms: Placebo (sugar pill)

SUMMARY:
Bupropion has been used successfully and safely for smoking cessation in adults. It was also used in very few studies among adolescent population. Our hypothesis is that Bupropion would be effective and safe among the adoelscent psychiatric population. A double-blind randomized controlled-trial will be held to determine that.

DETAILED DESCRIPTION:
The study will be conducted in Geha Mental Health Center. A total of 80 adolescent non-psychotic smokers will be recruited for this study. A smoker is defined as a cosumer of at least 5 cigarettes daily. A total of 80 patients will be recruited from the adolescent psychiatric wards or the adolescent clinics of the mental health center. The study group (N=40) will receive bupropion SR and the control group (N=40) will receive placebo medication. Age of participants will range from 13-20 years. Both genders will be included and all ethnic origins.

All participants will receive a detailed explanation about the study, its aims, the bupropion therapy, including possible adverse effects of the drug and other possible therapeutic alternatives. They will receive a leaflet summarizing all relevant data and information. Then they and their parents will sign an informed consent to participate in the study.

Procedure The mental health center's pharmacist will encapsulate the bupropion tablets, which will be supplied by the manufacturing company. The study capsules will all be kept in the hospital's pharmacy. Randomization will be performed using a random number table. The code will be held solely by the principal investigator, and will be broken in the end of the study's follow-up period, unless an emergency occurs. All participants will be given the telephone number of the principal investigator for any questions or problems arising.

The subjects in both groups will be double-blindly randomized to receive either bupropion or placebo. The assignment to each group will be done randomly in order to ensure location concealment. For subjects receiving bupropion, the dose will be 150 mg/d for the first three days, increasing for 150 mg twice daily, continued for a period of eight weeks. In case of intolerable side effects, the dosage will be decreased to 150 mg daily.

On recruitment, all subjects will be screened for-

* Medical history
* Vital signs
* Height
* Weight
* Place of birth
* Tobacco use history
* Alcohol and substance abuse
* Elctrocardiogram (ECG)
* Urine pregnancy test (for girls only)
* Kiddie schedule for affective disorders and schizophrenia (K-SADS-PL) screening tool (37).

Possible electrocardiographic side effects of bupropion that have been reported in the literature were tachycardia and conduction delays (widened QRS complex and/or prolonged QTc interval), but none of these delays progressed to a life-threatening arrhythmia, even in case of overdose.

Exclusion criteria will be:

* Psychiatric disorders in Axis I of DSM IV (38) (for the control group)
* Smoking less than 6 cigarettes a day
* Using other tobacco products other than cigarettes
* Using any other smoking cessation treatment
* Exhaled CO level of less than 10 ppm
* Convulsive disorder or a history of seizures
* A first-degree relative with a convulsive disorder
* Past sensitivity to bupropion.
* Positive pregnancy test
* lactation
* A lack of motivation to quit smoking
* Alcohol and substance abuse (or current alcohol withdrawal)
* Mental retardation and a lack of ability to give an informed consent
* Concurrent use of Monoamine oxidase inhibitors (MAO-I).
* Anorexia nervosa or bulimia nervosa.

All subjects will be evaluated for weight, smoking, substance use, anxiety and depressive symptoms at baseline, 1 month, 3 months, 6 months and 1 year. Follow-up phase will be blinded as well. Evaluation in these time points will include:

* Fagerstrom Tolerance Questionnaire modified for adolescents (FTQ( to measure nicotine dependence (39).
* Quantitive information on tobacco, alcohol and drug use (timeline followback methods)
* Children depression inventory (CDI) (40) to measure depression, translated and validated to hebrew (41).
* Children depression rating scale (CDRS) (42) to measure depression, translated and validated to hebrew (41)
* The Screen for Child Anxiety Related Emotional Disorders (SCARED) to measure anxiety (43;44)
* Exhaled air carbon monoxide (CO)
* Urine cotinine In addiction to the pharmacological therapy, both groups of the study will receive supportive and psychoeducational treatment in the setting of group therapy. Supportive psychotherapy focuses on using suggestions and supportive expressions to encourage the patient in his goal of quitting smoking. Psychoeducational treatment concentrates on educating the patients on the benefits of abandoning smoking and the use informative details in regards to that issue.

Main outcome measures: (1) Smoking cessation for 3 months. (2) Decrease in the carving to smoke.

ELIGIBILITY:
Inclusion Criteria:

* adolescents (age 13-20)
* daily smokers (over 5 cigarettes daily)
* have motivation to quit
* nonpsychotic
* treated in out MHC

Exclusion Criteria:

* Psychiatric disorders in Axis I of DSM IV (38) (for the control group)
* Smoking less than 6 cigarettes a day
* Using other tobacco products other than cigarettes
* Using any other smoking cessation treatment
* Exhaled CO level of less than 10 ppm
* Convulsive disorder or a history of seizures
* A first-degree relative with a convulsive disorder
* Past sensitivity to bupropion.
* Positive pregnancy test
* lactation
* A lack of motivation to quit smoking
* Alcohol and substance abuse (or current alcohol withdrawal)
* Mental retardation and a lack of ability to give an informed consent
* Concurrent use of Monoamine oxidase inhibitors (MAO-I).
* Anorexia nervosa or bulimia nervosa.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation | 3 months

SECONDARY OUTCOMES:
Decrease in craving | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Geha Mental Health Center, Petah Tikva, Israel

REFERENCES:
- [Background] Muramoto ML, Leischow SJ, Sherrill D, Matthews E, Strayer LJ. Randomized, double-blind, placebo-controlled trial of 2 dosages of sustained-release bupropion for adolescent smoking cessation. Arch Pediatr Adolesc Med. 2007 Nov;161(11):1068-74. doi: 10.1001/archpedi.161.11.1068. PMID 17984409